CLINICAL TRIAL: NCT02729818
Title: Adaptation Time Required for the Optimisation of Maia Microperimetry Visual Field Testing
Status: Completed | Type: Observational
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Other Study IDs: DarkAdapt
Record Dates: First submitted 2016-02-25; First posted 2016-04-06 (Estimated); Last update posted 2018-11-08 (Actual); Status verified 2017-10

CONDITIONS: Retina; Change
Keywords: Retina; Microperimetry; Visual Fields

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Microperimetry is a relatively new and extremely sensitive method of assessing visual function. It projects light stimuli onto a defined area of the retina to map retinal perceptual thresholds. Participants look at a focal point and press a button to indicate when they have seen a light stimulus. The stimuli vary in intensity to find the participant's visual sensitivity.

Microperimetry is carried out in low light conditions. Before testing, participants must adapt to the low light conditions in a process called 'dark adaptation.' Currently there is no consensus on the optimal time needed for dark adaptation. Investigators know that visual sensitivity differs in differing light conditions. Failing to sufficiently dark-adapt may therefore adversely affect test results.

The aim of this study is to establish the optimal length of dark adaptation for microperimetry performance in healthy volunteers. On day 1, participants will undergo training field tests to reduce a learning effect affecting the results. Tests will then be performed following 5 mins adaptation, 10 mins adaptation and 30mins adaptation, On day 2, participants will perform testing following no adaptation time, 15 mins adaptation, and 20 mins adaptation. Statistics will be used to determine the effect of adaptation time on average threshold measures.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study.
* Male or female.
* Age 18 - 60 years.
* Best corrected visual acuity of at least Logmar 0.1 in right eye.
* Able to tolerate physical requirements of microperimetry testing i.e. able to sit still at the microperimeter in dark environment and indicate when a light stimulus has been seen using the provided button.

Exclusion Criteria:

* Any co-existing ocular pathology, either pre-existing or identified on initial ocular examination, not including refractive error or previous cataract surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Forty healthy adult volunteers (over 18) will be recruited from the University of Oxford. They will need to have healthy eyes and good eyesight (better than 6/7.5 Snellen visual acuity), with no eye diseases apart from refractive error (needing to wear glasses or contact lenses). Participants will need to be able to sit upright at the microperimeter (which involves putting their chin on a chin rest and being able to sit still for up to 20 minutes at a time), and be able to press a button to indicate when they have seen a light stimulus.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Change in average threshold of tests following different dark adaptation periods will be compared. | Different time intervals for adaptation prior to testing; 0 minutes, 5, 10, 15, 20 and 30 minutes on day 1 and day 2.
  The average threshold for each test is detailed on the microperimetry printout and is measured in dB. This will be measured by testing following each time interval specified.

SECONDARY OUTCOMES:
Change in fixation stability, as defined by the area in which 95% of the fixation points for any specific test fall, following different dark adaptation periods will be compared. | Different time intervals for adaptation prior to testing; 0 minutes, 5, 10, 15, 20 and 30 minutes on day 1 and day 2
  The fixation stability for each test is detailed on the microperimetry printout and is measured in degrees for the area covering 95% of the fixation points. This will be measured by testing following each time interval specified.

CONTACTS AND LOCATIONS:
Overall Officials: Jasleen K Jolly, Principal Investigator — University of Oxford
Locations (1):
- Nuffield Laboratory of Ophthalmology, Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Han RC, Gray JM, Han J, Maclaren RE, Jolly JK. Optimisation of dark adaptation time required for mesopic microperimetry. Br J Ophthalmol. 2019 Aug;103(8):1092-1098. doi: 10.1136/bjophthalmol-2018-312253. Epub 2018 Sep 29. PMID 30269100
- See also: Related Info — https://www.ndcn.ox.ac.uk/divisions/nlo/